CLINICAL TRIAL: NCT02555696
Title: Assessment of Abraxane in Metastatic Breast Cancer in a Real-life Setting
Brief Title: Abraxane in Treatment of Metastatic Breast Cancer
Status: Completed | Type: Observational
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: NIPMS-Celgene-AUT-002
Record Dates: First submitted 2015-09-18; First posted 2015-09-21 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic Breast Cancer; nab-paclitaxel; Abraxane
MeSH Terms: conditions — Breast Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- nab-paclitaxel: nab-paclitaxel 260mg/m^2 in intravenous (IV) infusion every 3 weeks until progression or toxicity
  Interventions: Drug: nab-paclitaxel

INTERVENTIONS:
Drug: nab-paclitaxel — nab-paclitaxel by IV infusion every 3 weeks until progression or toxicity
  Other Names: Abraxane; ABI-007

SUMMARY:
This observational project is collecting tolerability, safety and efficacy data with the routine use of Abraxane in the treatment of metastatic breast cancer. Additionally data on the dosage of Abraxane and general data on the disease and the health status of the patient will be collected.

DETAILED DESCRIPTION:
This observational program is aimed at gaining tolerability, safety and efficacy data with the routine use of Abraxane in its labelled indication in metastatic breast cancer. Additionally data on real life dosing in daily clinical routine will be analyzed.

A detailed record of the medical history including co-morbidities and pre-treatment regimens will allow analysis of the impact thereof on tolerability, dosage and efficacy.

This data might also be supportive for further treatment optimization of Abraxane in Metastatic Breast Cancer (MBC).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with metastatic breast cancer (according to European Summary of Product characteristics (SmPC)
2. Signed Informed Consent
3. Participants > 18 Years of Age

Exclusion Criteria:

1. Pregnant or lactating females
2. Neutrophils <1.5 X 10^9/L
3. Hypersensivity to nab-paclitaxel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2012-05-31 (Actual); Primary Completion 2016-02-28 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Up to 3 years
  Includes the number of participants with adverse events

SECONDARY OUTCOMES:
Overall Response | Up to 3 years
  Number of participants who achieve a response

CONTACTS AND LOCATIONS:
Overall Officials: Guenter Voraberger, Study Chair — Celgene
Locations (13):
- Austria (13):
  - LKH Feldkirch, Feldkirch
  - Medical University Graz, Graz
  - Medical University Innsbruck, Innsbruck
  - LKH Leoben, Leoben
  - KH Barmherzige Schwestern Linz, Linz
  - LKH Salzburg, Salzburg
  - LKH St. Pölten, Sankt Pölten
  - LKH Steyr, Steyr
  - Medical University Vienna, Vienna
  - KH SMZ Ost, Vienna
  - LKH Vöcklabruck, Vöcklabruck
  - Klinikum Wels, Wels
  - LKH Wr. Neustadt, Wiener Neustadt